CLINICAL TRIAL: NCT01273571
Title: An Open-Label, Fixed Sequence Study to Investigate the Potential for Pharmacokinetic and Pharmacodynamic Interaction Between Single-Dose Metformin and Multiple-Dose Canagliflozin in Healthy Subjects
Brief Title: A Pharmacokinetic and Pharmacodynamic Study of Metformin and Canagliflozin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017815; 28431754DIA1028
Record Dates: First submitted 2010-12-23; First posted 2011-01-10 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Canagliflozin; Metformin (GLUCOPHAGE IR); Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Canagliflozin; Metformin

ARMS (1):
- 001 (Experimental): Canagliflozin/Metformin Two 1000-mg tablets of metformin on Day 1 followed by one 300-mg tablet of canagliflozin once daily on Days 4 through 8 followed by two 1000-mg tablets of metformin and one 300-mg tablet of canagliflozin on Day 8.
  Interventions: Drug: Canagliflozin/Metformin

INTERVENTIONS:
Drug: Canagliflozin/Metformin — Two 1000-mg tablets of metformin on Day 1 followed by one 300-mg tablet of canagliflozin once daily on Days 4 through 8, followed by two 1000-mg tablets of metformin and one 300-mg tablet of canagliflozin on Day 8.

SUMMARY:
The purpose of the study is to investigate the potential interaction between multiple oral doses of canagliflozin and a single oral dose of metformin in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center study of canagliflozin and metformin in healthy adult volunteers. Canagliflozin (a Sodium-Glucose Cotransporter 2 inhibitor) is currently under development to lower blood sugar levels in patients with type 2 diabetes mellitus (T2DM) and metformin is an approved treatment for patients with T2DM. Canagliflozin will be administered orally (by mouth) as a single 300-mg tablet on Days 4, 5, 6, 7, and 8 and metformin will be administered orally as two 1,000 mg tablets on Days 1 and 8. Both canagliflozin and metformin tablets will be taken with 8 ounces (240 mL) of water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 18 and 30 kg/m2, inclusive.

Exclusion Criteria:

* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to canagliflozin or metformin or any of the excipients of the formulation of canagliflozin or metformin
* Known allergy to heparin or history of heparin induced thrombocytopenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin | At protocol-specified times up to Day 11
Plasma concentrations of metformin | At protocol-specified times up to Day 11)
Urine concentrations of metformin | At protocol-specified times up to Day 10)
Plasma concentrations of glucose | Up to Day 9
Urinary glucose excretion (UGE) | Up to Day 11

SECONDARY OUTCOMES:
The number and type of adverse events reported | Up to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Murphy J, Skee D, Wajs E, Mamidi RN, Tian H, Vandebosch A, Wang SS, Verhaeghe T, Stieltjes H, Usiskin K. Effect of canagliflozin on the pharmacokinetics of glyburide, metformin, and simvastatin in healthy participants. Clin Pharmacol Drug Dev. 2015 May-Jun;4(3):226-36. doi: 10.1002/cpdd.166. Epub 2014 Oct 27. PMID 27140803